CLINICAL TRIAL: NCT01814956
Title: Prospective, Randomized, Controlled, Double-blind, Parallel-group, Mono-center, Explorative Phase IV Trial on the Efficacy and Safety of a Fish Oil Containing Lipid Emulsion Versus a Standard Soybean-oil Based Lipid Emulsion in Patients With Acute Lung Injury
Brief Title: Different Lipid Emulsions in Acute Lung Injury Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-0813; 2011-003397-82 (EudraCT Number)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): i.v. lipid emulsion for parenteral nutrition
  Interventions: Drug: Lipoplus 20%
- 2 (Active Comparator): i.v. lipid emulsion for parenteral nutrition
  Interventions: Drug: Lipofundin N 20%

INTERVENTIONS:
Drug: Lipoplus 20% — Lipoplus 20% (MCT/LCT/FO) i.v. lipid emulsion for parenteral nutrition
  Arms: 1
Drug: Lipofundin N 20% — Lipofundin N 20% (LCT, soy bean oil) i.v. lipid emulsion for parenteral nutrition
  Arms: 2

SUMMARY:
Aim is to investigate the influence of an early supply of parenteral nutrition including a fish oil containing lipid emulsion on the course of acute lung injury in the intensive care unit. In comparison, a standard parenteral nutrition with a soybean oil based emulsion will be used. Data obtained in this trial may provide evidence for a beneficial effect of fish oil derived omega-3 fatty acids in parenteral nutrition regarding their influence on acute lung injury.

ELIGIBILITY:
Inclusion:

* Acute Lung Injury as a result of proven pneumonia (x-ray) or witnessed aspiration
* Oxygenation factor ≤ 300
* <= 72 hours since intubation or non-invasive ventilatory support by mask at screening
* Expected need for parenteral nutrition for at least 5 days
* Male or female ≥ 18 years of age

Exclusion:

* Exclusion of pregnancy in women with child-bearing potential
* Cardiogenic pulmonary oedema
* Previous (< 1 month) or ongoing need for corticosteroids >0.1 mg/kg/d prednisolon-equivalent or other immune suppressive treatment
* Active or previous (< 1 year) treatment for solid or haematologic malignancy
* Serum triglycerides > 300 mg/dl at screening
* Alterations of coagulation (thrombocytes <100 Giga/l), aPTT > 60 sec, INR ≥ 2.5 without therapeutic intervention
* Autoimmune disease or HIV (according to medical history)
* Known or suspected drug abuse
* General contraindications to infusion therapy :

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
change in blood oxygenation (PaO2/FiO2ratio) | change day 1 to day 6

SECONDARY OUTCOMES:
Triglycerides | day 1 to day 16
Sequential Organ Failure Assessment | day 1 to day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Giessen, Giessen, Germany